CLINICAL TRIAL: NCT05406986
Title: The Effect of Care Bundle in Preventing Pressure Ulcers Caused by Medical Devices in the Pediatric Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, Erhan Elmaoğlu, research assistant, Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Kilis7AralikUnivesity2022
Record Dates: First submitted 2022-04-24; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Pressure Ulcer; Nursing Caries; Device Induced Injury
Keywords: medical devices; pressure ulcers; Care Bundles
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Experimental and control groups will be selected using the randomized control method.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group to which the care bundle will be applied (Experimental): Patients with a score of 13 or higher on the Braden QD medical instrument risk assessment scale.
  Patients with attached nasogastric tube, intubation tube and saturation probe.
  Interventions: Other: care bundle application
- group not to be interfered with (No Intervention): Patients with attached nasogastric tube, intubation tube and saturation probe.

INTERVENTIONS:
Other: care bundle application — The patients in the experimental group will be given care according to the current care bundle for 14 days
  Arms: the group to which the care bundle will be applied

SUMMARY:
With the development of technology in medicine, more medical instruments are used in the treatment of diseases. Although the use of these instruments provides great benefits for the patients, it can also cause some complications.One of the most important of these complications is pressure ulcer.Some care and evaluation are needed to prevent these complications.This study aims to prevent pressure ulcers with a care package for patients with high risk scores.

DETAILED DESCRIPTION:
A care package will be created with the Delphi method to prevent pressure ulcers caused by medical devices.Experimental and control groups will be formed by randomized control method.The care package created for 14 days will be applied to the experimental group. standard care will be applied to the control group.As a result, the rates of medical device-induced pressure ulcers in both groups will be compared.Children between the ages of 1 and 10 years and treated in the pediatric intensive care unit will be included in the study.Patients with any skin-related disease will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* being in the pediatric intensive care unit.
* nasogastric tube, intubation tube and saturation probe attached.
* Voluntary consent of family to participate in the study

Exclusion Criteria:

* Patients with skin disease
* Patients staying less than 14 days

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer | 14 day
  Medical devices related pressure ulcer

SECONDARY OUTCOMES:
medical device induced pressure ulcer | 14 day
  The rate of pressure ulcers caused by medical devices in the care package group will be compared with the rates of pressure ulcers caused by medical devices in patients receiving normal care.

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin Çiğdem, Principal Investigator — Hasan Kalyoncu Univesity

IPD SHARING:
Plan to Share IPD: No
The data collected by the researcher will be shared with other participants. however, information about the patient will not be shared.

REFERENCES:
- [Result] Butler CT. Pediatric skin care: guidelines for assessment, prevention, and treatment. Dermatol Nurs. 2007 Oct;19(5):471-2, 477-82, 485. PMID 18286861
- [Result] Curley MAQ, Hasbani NR, Quigley SM, Stellar JJ, Pasek TA, Shelley SS, Kulik LA, Chamblee TB, Dilloway MA, Caillouette CN, McCabe MA, Wypij D. Predicting Pressure Injury Risk in Pediatric Patients: The Braden QD Scale. J Pediatr. 2018 Jan;192:189-195.e2. doi: 10.1016/j.jpeds.2017.09.045. PMID 29246340
- [Result] Freundlich K. Pressure Injuries in Medically Complex Children: A Review. Children (Basel). 2017 Apr 7;4(4):25. doi: 10.3390/children4040025. PMID 28387749
- [Result] Puspitasari JD, Nurhaeni N, Waluyanti FT. Testing of Braden QD Scale for predicting pressure ulcer risk in the Pediatric Intensive Care Unit. Pediatr Rep. 2020 Jun 25;12(Suppl 1):8694. doi: 10.4081/pr.2020.8694. eCollection 2020 Jun 25. PMID 32904968
- [Result] Delmore BA, Ayello EA. CE: Pressure Injuries Caused by Medical Devices and Other Objects: A Clinical Update. Am J Nurs. 2017 Dec;117(12):36-45. doi: 10.1097/01.NAJ.0000527460.93222.31. PMID 29120893